CLINICAL TRIAL: NCT02275234
Title: A Feasibility Study of Implementing a Simple Psychological Intervention in Survivors of Cardiac Arrest and Their Family Members/Friend to Assess the Impact on Their Quality of Life and Cognitive Function
Brief Title: Care After Resuscitation
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: B709
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; psychological intervention
MeSH Terms: conditions — Heart Arrest | interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Patients who survived cardiac arrest >3 months prior to the start of the study and a close family/friend,will be invited to attend an outpatient clinic
- Prospective- psychological intervention: In patients who survived cardiac arrest and a close family/friend,will be invited to attend an outpatient clinic
  Interventions: Other: Psychological intervention

INTERVENTIONS:
Other: Psychological intervention — Psychological support via clinic visit, helpline and telephone calls
  Groups: Prospective- psychological intervention

SUMMARY:
The purpose of this study is to investigate whether simple psychological interventions can be implemented at the Essex Cardiothoracic Centre (CTC) with a view to supporting the psychological wellbeing of survivors of cardiac arrest during their recovery.

DETAILED DESCRIPTION:
At the Essex Cardiothoracic Centre (CTC) the follow up of patients surviving cardiac arrest demonstrated that standard psychological support arrangements for patients and their families/relatives were inadequate.

The purpose of this study is to investigate simple psychological interventions can be implemented here at the Essex CTC with a view to supporting the psychological wellbeing of survivors of cardiac arrest during their recovery.

The investigators propose to recruit 2 groups of patients. The first group will be chosen from patients who have already survived a cardiac arrest > 3 months prior to the start of the study. Participants in this group (patient and a relative/friend) will be invited to attend an outpatient clinic at the Essex CTC with members of the research team. The investigators will record general physical health condition and psychological wellbeing, using recommended questionnaires. A referral to onsite consultant psychiatrist will be offered to anyone expressing signs of severe depression.

The second group will be recruited from patients who survive cardiac arrest from the start of study date. Participants in this group (patient and a relative/friend) will be approached by a member of the research team whilst in hospital and an informed consent will be obtained. Baseline data will be acquired using the recommended questionnaires and a supportive psychological intervention will be offered in the form of a dedicated telephone helpline, attendance at a cardiac arrest clinic and early referral to clinical psychiatrist if appropriate for psychological help. At around 6 months from the date of cardiac arrest, participants will be invited to attend a clinic to reevaluate post cardiac arrest care using the same recommended questionnaires. At the end of the study, the data between the 2 groups will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Anyone surviving cardiac arrest
* Age greater than or equal to 18 yrs
* Cerebral Performance Category (CPC) 1-2 at the time of discharge from hospital
* English speaking
* Able to give informed consent

Exclusion Criteria:

* Age less than 18yrs
* CPC 3-5 at the time of discharge from hospital
* Non-English speaking
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective and prospective cohort of patients following cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by responses on SF36 | 6 months
  Change in Quality of Life before and after psychological intervention in patients surviving cardiac arrest and their family/friends
Change in cognitive function as measured by responses on Montreal Cognitive function tool | 6 months
  Change in cognitive function before and after psychological intervention in patients surviving cardiac arrest and their family/friends
Change in cognitive function as measured by responses on Cogfail questionnaire | 6 months
  Change in cognitive function before and after psychological intervention in patients surviving cardiac arrest and their family/friends

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Keeble, MBBS MD MRCP, Principal Investigator — Basildon and Thurrock University Hospitals NHS FT
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No